CLINICAL TRIAL: NCT05034952
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Multi-dose Study Evaluating the Efficacy and Safety of VX-548 for Acute Pain After an Abdominoplasty
Brief Title: A Study Evaluating Efficacy and Safety of VX-548 for Acute Pain After an Abdominoplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX21-548-102
Record Dates: First submitted 2021-08-27; First posted 2021-09-05 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Participants received placebo matched to VX-548 and Hydrocodone bitartrate/ acetaminophen (HB/APAP) for 2 days.
  Interventions: Drug: Placebo (matched to VX-548); Drug: Placebo (matched to HB/APAP)
- HB/APAP (Active Comparator): Participants received HB 5 mg / APAP 325 milligrams (mg) every 6 hours (q6h) for 2 days.
  Interventions: Drug: HB/APAP
- VX-548: Low Dose (Experimental): Participants received VX-548 60 mg as first dose, followed by VX-548 30 mg every 12 hours (q12h) for 2 days.
  Interventions: Drug: VX-548
- VX-548: High Dose (Experimental): Participants received VX-548 100 mg as first dose, followed by VX-548 50 mg q12h for 2 days.
  Interventions: Drug: VX-548

INTERVENTIONS:
Drug: VX-548 — Tablets for oral administration.
  Other Names: Suzetrigine
  Arms: VX-548: High Dose; VX-548: Low Dose
Drug: HB/APAP — Capsules for oral administration.
  Arms: HB/APAP
Drug: Placebo (matched to VX-548) — Placebo matched to VX-548 for oral administration.
  Arms: Placebo
Drug: Placebo (matched to HB/APAP) — Placebo matched to HB/APAP for oral administration.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of VX-548 doses in treating acute pain after an abdominoplasty.

ELIGIBILITY:
Key Inclusion Criteria:

* Before Surgery:

  * Participant scheduled to undergo an abdominoplasty without collateral procedures
* After Surgery:

  * Participant is lucid and able to follow commands
  * All analgesic guidelines were followed during and after the abdominoplasty
  * Abdominoplasty procedure duration <=3 hours without collateral procedures (for example., liposuction)

Key Exclusion Criteria

* Before Surgery:

  * Prior history of abdominoplasty, intra-abdominal and/or pelvic surgery
  * History of cardiac dysrhythmias requiring anti-arrhythmia treatment(s)
  * Any prior surgery within 1 month before the first study drug
* After Surgery:

  * Participant had medical complications during the abdominoplasty that, in the opinion of the investigator, should preclude randomization
  * Participant had collateral procedures during the abdominoplasty

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2021-12-05 (Actual); Study Completion 2021-12-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Arizona Research Center, Phoenix, Arizona
  - Lotus Clinical Research, Pasadena, California
  - Chesapeake Research Group, Pasadena, Maryland
  - Midwest Clinical Research Center, Dayton, Ohio
  - First Surgical Hospital, Bellaire, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - JBR Clinical Research, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing

REFERENCES:
- [Derived] Jones J, Correll DJ, Lechner SM, Jazic I, Miao X, Shaw D, Simard C, Osteen JD, Hare B, Beaton A, Bertoch T, Buvanendran A, Habib AS, Pizzi LJ, Pollak RA, Weiner SG, Bozic C, Negulescu P, White PF; VX21-548-101 and VX21-548-102 Trial Groups. Selective Inhibition of NaV1.8 with VX-548 for Acute Pain. N Engl J Med. 2023 Aug 3;389(5):393-405. doi: 10.1056/NEJMoa2209870. PMID 37530822

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebos matched to VX-548 and Hydrocodone bitartrate/acetaminophen (HB/APAP) for 2 days.
- HB/APAP: Participants received HB 5 milligrams (mg) / APAP 325 mg every 6 hours for 2 days.
Period: Overall Study
Arm/Group | Placebo | HB/APAP | VX-548: Low Dose | VX-548: High Dose
Started | 77 | 76 | 74 | 76
Completed | 75 | 70 | 70 | 72
Not Completed | 2 | 6 | 4 | 4
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Withdrawal of consent (not due to AE) | 0 | 2 | 1 | 0
Not completed — Lost to Follow-up | 1 | 4 | 3 | 3
Not completed — Other | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who had received at least one dose of the study drug during the treatment period were included in the baseline analysis.
Groups:
- Placebo: Participants received placebo matched to VX-548 and HB/APAP for 2 days.
- HB/APAP: Participants received HB 5 mg / APAP 325 mg q6h for 2 days.
- VX-548: Low Dose: Participants received VX-548 60 mg as first dose, followed by VX-548 30 mg q12h for 2 days.
- Total: Total of all reporting groups
Arm/Group | Placebo | HB/APAP | VX-548: Low Dose | VX-548: High Dose | Total
Number analyzed (Participants) | 77 | 76 | 74 | 76 | 303
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (9.5) | 45.4 (10.7) | 41.5 (9.2) | 43.1 (9.7) | 43.2 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 73 | 74 | 75 | 298
  Male | 1 | 3 | 0 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 20 | 21 | 25 | 80
  Not Hispanic or Latino | 63 | 56 | 53 | 51 | 223
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 57 | 53 | 57 | 57 | 224
  Black or African American | 20 | 18 | 15 | 13 | 66
  American Indian or Alaska Native | 0 | 1 | 0 | 1 | 2
  Native Hawaiian or other Pacific Islander | 0 | 2 | 0 | 2 | 4
  Other | 0 | 2 | 1 | 1 | 4
  Multiracial | 0 | 0 | 1 | 2 | 3
Pain Intensity at Baseline (at 0 hours) as Recorded on Numeric Pain Rating Scale (NPRS) [Mean (Standard Deviation); unit: units on a scale] — Pain intensity was recorded on 11-point NPRS, score range: 0 to 10, where 0=no pain and 10=worst imaginable pain.
  units on a scale | 7.4 (1.6) | 7.3 (1.8) | 7.4 (1.8) | 7.2 (1.7) | 7.3 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Time-weighted Sum of the Pain Intensity Difference (SPID) as Recorded on a Numeric Pain Rating Scale (NPRS) at Rest 0 to 48 Hours (SPIDr0-48) After the First Dose of Study Drug
Description: SPID was calculated as the sum of the product of time (in hours) elapsed since previous measurements and pain intensity difference. Pain intensity difference was calculated by subtracting the pain intensity score at given post-dose time points from the baseline pain intensity scores (using pain rating score range: 0= no pain to 10= worst possible pain). SPIDr0-48 was calculated from 0 to 48 hours and the score range was -480 (worst score) to 480 (best score).
Time Frame: 0 to 48 Hours After First Dose of Study Drug
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | HB/APAP | VX-548: Low Dose | VX-548: High Dose
Number analyzed (Participants) | 77 | 76 | 74 | 76
units on a scale | 72.73 (10.23) | 85.20 (10.30) | 95.11 (10.44) | 110.53 (10.30)
Statistical Analysis 1: Comparison: Placebo vs HB/APAP; Test type: Superiority; p = 0.3914, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs VX-548: Low Dose; Test type: Superiority; p = 0.1266, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs VX-548: High Dose; Test type: Superiority; p = 0.0097, ANCOVA

2. Secondary Outcome: Time-weighted SPID as Recorded on an NPRS at Rest 0 to 24 Hours (SPIDr0-24) After the First Dose of Study Drug
Description: SPID was calculated as the sum of the product of time (in hours) elapsed since previous measurements and pain intensity difference. Pain intensity difference was calculated by subtracting the pain intensity score at given post-dose time points from the baseline pain intensity scores (using pain rating score range: 0= no pain to 10= worst possible pain). SPIDr0-24 was calculated from 0 to 24 hours and the score range was -240 (worst score) to 240 (best score).
Time Frame: 0 to 24 Hours After First Dose of Study Drug
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | HB/APAP | VX-548: Low Dose | VX-548: High Dose
Number analyzed (Participants) | 77 | 76 | 74 | 76
units on a scale | 25.96 (4.70) | 29.98 (4.73) | 37.65 (4.79) | 45.54 (4.73)
Statistical Analysis 1: Comparison: Placebo vs HB/APAP; Test type: Superiority; p = 0.5476, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs VX-548: Low Dose; Test type: Superiority; p = 0.0825, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs VX-548: High Dose; Test type: Superiority; p = 0.0036, ANCOVA

3. Secondary Outcome: Percentage of Participants With at Least 30 Percent (%),Reduction in NPRS (at Rest) at 48 Hours After the First Dose of Study Drug
Description: Pain intensity was recorded on 11-point NPRS, score range: 0 to 10, where 0= no pain and 10= worst imaginable pain. The percentage of participants with at least 30% reduction from baseline in NPRS at 48 hours after the first dose of VX-548 or placebo were reported.
Time Frame: From Baseline At 48 Hours After First Dose of Study Drug
Population: FAS.
Measure: Number; unit: percentage of participants
Groups:
- HB/APAP: Participants received HB 5 mg/APAP 325 mg q6h for 2 days.
Arm/Group | Placebo | HB/APAP | VX-548: Low Dose | VX-548: High Dose
Number analyzed (Participants) | 77 | 76 | 74 | 76
percentage of participants | 48.1 | 53.9 | 59.5 | 60.5
Statistical Analysis 1: Comparison: Placebo vs HB/APAP; Test type: Superiority; p = 0.4712, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs VX-548: Low Dose; Test type: Superiority; p = 0.1635, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs VX-548: High Dose; Test type: Superiority; p = 0.1158, Cochran-Mantel-Haenszel

4. Secondary Outcome: Percentage of Participants With at Least 50% Reduction in NPRS (at Rest) at 48 Hours After the First Dose of Study Drug
Description: Pain intensity was recorded on 11-point NPRS, score range: 0 to 10, where 0=no pain and 10=worst imaginable pain. The percentage of participants with at least 50% reduction from baseline in NPRS at 48 hours after the first dose of VX-548, HB/APAP, or placebo were reported.
Time Frame: From Baseline At 48 Hours After First Dose of Study Drug
Population: FAS.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | HB/APAP | VX-548: Low Dose | VX-548: High Dose
Number analyzed (Participants) | 77 | 76 | 74 | 76
percentage of participants | 33.8 | 42.1 | 43.2 | 44.7
Statistical Analysis 1: Comparison: Placebo vs HB/APAP; Test type: Superiority; p = 0.2882, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs VX-548: Low Dose; Test type: Superiority; p = 0.2344, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs VX-548: High Dose; Test type: Superiority; p = 0.1724, Cochran-Mantel-Haenszel

5. Secondary Outcome: Percentage of Participants With at Least 70% Reduction in NPRS (at Rest) at 48 Hours After the First Dose of Study Drug
Description: Pain intensity was recorded on 11-point NPRS, score range: 0 to 10, where 0= no pain and 10= worst imaginable pain. The percentage of participants with at least 70% reduction from baseline in NPRS at 48 hours after the first dose of VX-548,HB/APAP or placebo were reported.
Time Frame: From Baseline at 48 Hours After First Dose of Study Drug
Population: FAS.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Participants received placebos matched to VX-548 and HB/APAP for 2 days.
Arm/Group | Placebo | HB/APAP | VX-548: Low Dose | VX-548: High Dose
Number analyzed (Participants) | 77 | 76 | 74 | 76
percentage of participants | 14.3 | 23.7 | 18.9 | 25.0
Statistical Analysis 1: Comparison: Placebo vs HB/APAP; Test type: Superiority; p = 0.1343, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs VX-548: Low Dose; Test type: Superiority; p = 0.4501, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs VX-548: High Dose; Test type: Superiority; p = 0.1009, Cochran-Mantel-Haenszel

6. Secondary Outcome: Safety and Tolerability as Assessed by Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Day 16
Population: Safety set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- HB/APAP: Participants received HB 5 mg / APAP 325 mg every 6 hours for 2 days.
Arm/Group | Placebo | HB/APAP | VX-548: Low Dose | VX-548: High Dose
Number analyzed (Participants) | 77 | 76 | 74 | 76
Participants
  Participants with TEAEs | 54 | 46 | 45 | 42
  Participants with SAEs | 1 | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 16
Groups:
- VX-548 Low Dose: Participants received VX-548 60 mg as first dose, followed by VX-548 30 mg q12h for 2 days.
- VX-548 High Dose: Participants received VX-548 100 mg as first dose, followed by VX-548 50 mg q12h for 2 days.
Arm/Group | Placebo | HB/APAP | VX-548 Low Dose | VX-548 High Dose
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/76 | 0/74 | 0/76
Serious Adverse Events (participants affected / at risk) | 1/77 | 1/76 | 1/74 | 0/76
Other Adverse Events (participants affected / at risk) | 40/77 | 37/76 | 37/74 | 33/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=77) | HB/APAP (N=76) | VX-548 Low Dose (N=74) | VX-548 High Dose (N=76)
Incision site cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=77) | HB/APAP (N=76) | VX-548 Low Dose (N=74) | VX-548 High Dose (N=76)
Constipation (Gastrointestinal disorders) | 4 | 9 | 7 | 7
Nausea (Gastrointestinal disorders) | 28 | 23 | 22 | 14
Vomiting (Gastrointestinal disorders) | 5 | 8 | 1 | 2
Dizziness (Nervous system disorders) | 14 | 8 | 11 | 6
Headache (Nervous system disorders) | 5 | 5 | 6 | 11
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 2 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 2 | 4 | 1
Hypotension (Vascular disorders) | 3 | 3 | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-01-21): https://cdn.clinicaltrials.gov/large-docs/52/NCT05034952/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/52/NCT05034952/SAP_001.pdf